CLINICAL TRIAL: NCT00765791
Title: 2B or Not 2B? Shoulder Function After Level 2B Neck Dissection: A Randomized Controlled
Brief Title: 2B or Not 2B? Shoulder Function After Level 2B Neck Dissection: A Randomized Controlled Study
Acronym: 2BN2B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7527
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2019-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck cancer; oral cancer; oropharyngeal cancer; laryngeal cancer; selective neck dissection; submuscular recess; level 2b
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Mouth Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Not 2B) (Active Comparator): Selective neck dissection is performed on the dominant arm. Level 2B is not dissected.
  Interventions: Procedure: Selective Neck Dissection Excluding Level 2B
- Group 2 (2B) (Active Comparator): Selective neck dissection is performed on the dominant arm. Level 2B is dissected.
  Interventions: Procedure: Selective Neck Dissection Including Level 2B

INTERVENTIONS:
Procedure: Selective Neck Dissection Excluding Level 2B — Selective neck dissection is performed. Level 2a is dissected; level 2b is not dissected.
  Other Names: Not 2B
  Arms: Group 1 (Not 2B)
Procedure: Selective Neck Dissection Including Level 2B — Selective neck dissection is performed. Level 2a is dissected; level 2b is also dissected.
  Other Names: 2B
  Arms: Group 2 (2B)

SUMMARY:
Many types of head and neck cancers will have local spread to the neck. As such selective neck dissection is performed as part of the treatment. The neck is divided into various levels. Selective neck dissection targets areas that are most likely to harbor cancer cells for specific types of head and neck cancers. Level IIB has been particularly controversial in the last few years, as the rate of cancer spread to this area has been shown to be quite low (0-8%). Moreover, because the spinal accessory nerve (involved in shoulder function) runs through this area, there is theoretical risk of causing post-operative shoulder weakness. As such, the question of whether removing level IIB, knowing that there is low chance of it containing disease spread, is worth risking decreased shoulder function. Some would argue that all potential diseased sites should be removed at all costs. While other advocate that a balance between disease cure and function should be maintained. However, what needs to be determined is just what impact does dissecting IIB have on shoulder function. At our institution, the rate of poor shoulder function associated with selective neck dissection has been perceived as being quite low. This study is designed to test this observation.

Hypothesis: Neck dissection including level IIb in head and neck cancer patients will not lead to worse shoulder function and quality of life than when level IIb is preserved.

DETAILED DESCRIPTION:
The lymphatic fluid of upper aerodigestive tract (UADT) drains into various levels of the neck. When cancer occurs in the UADT, the potential for local metastatic spread to the neck exists, thus necessitating treatment of the neck. Ideally all potential neck structures, which could harbor cancer cells or provide a dock for recurrence, would be eradicated. Unfortunately, such radical treatments have shown to cause extreme rates of morbidity with little extra oncologic benefit. Thus, head and neck oncologists have strived to create treatment paradigms, which maximize cure rates while minimizing morbidity. Finding this intricate balance has translated to selective neck dissection (SND) and post-operative RT.1

Increased understanding of lymphatic drainage patterns in the head and neck has lead to widespread use of SND. Through removal of lymphatics in neck levels with the highest risk of harboring cancer cells, based on primary tumor site, important neck structures may be preserved. As such, the treatment remains oncologically sound and avoids the morbidity associated with its predecessor, the radical neck dissection. 1

One of the structures preserved in the SND is the spinal accessory nerve (SAN), which is responsible for providing motor innervation to the sternocleidomastoid (SCM) and trapezius muscles. Thus, it is intricately involved in shoulder function. The nerve exists the skull base at the jugular foramen and obliquely passes through neck level II. It then passes posterior to the SCM and eventually enters the trapezius muscles. Through this trajectory, it divides level II into IIa (anterior to the SAN) and IIb (posterior to the SAN).

It is known that shoulder function significantly deteriorates when level V is dissected.2 This is likely due to traction and devascularization injury of the longest portion of the SAN in the neck. As such, practice has become such that level V is left intact in cases where it does not harbor detectable disease or when occult disease incidence is very low. Due to the intimate relationship of IIb with the SAN, there is also potential for injury to the nerve in this area.2 As such, debate has arisen to the necessity of including IIb in the neck dissection specimen. Studies have shown that the prevalence of occult nodal disease in IIb ranges from 0-8.7.5% depending on the overall n stage of the neck.3-5 These figures have lead head and neck surgeons to weigh the benefits of not excising lymphatic tissue with low nodal metastatic rates versus excising the area and decreasing post-operative shoulder function.6

Because the incidence of occult metastases in IIb is low3-5, it has become standard of care in many centers to spare IIb, if it is oncologically feasible, in SND to preserve shoulder function. Because these patients receive post-operative RT it is thought that the RT will address any occult disease. Unfortunately, relying on RT poses two problems:

1. occult disease may not respond to the RT
2. leaving level IIb intact provides a lymphatic route of recurrence despite undergoing RT By surgically removing all portals of lymphatic disease spread these issues above can be eliminated.

The goal of this study is to demonstrate that the minimal manipulation of the SAN associated with IIb dissection will not have a significant impact on post-operative shoulder function. If this is the case, the standard of practice should be changed to include IIb in the SND specimen in cases where level IIa is dissected as well. This would eliminate any further lymphatic tissue, which may harbor disease.

Note: At the University of Alberta, some head and neck surgeons prefer to spare IIb in SND, while others prefer to resect it. Thus, the protocol in this study does not manipulate current standards of practice.

*Reference numbers correspond to articles in the "Citations" section. The citations are in order of appearance in the above text.

ELIGIBILITY:
Inclusion Criteria:

1. Head and neck cancer to be treated with primary surgical resection, SND and post-operative radiation therapy (RT).
2. N0 neck disease on side of the dominant hand
3. Willingness to participate in post-operative physiotherapy

Exclusion Criteria:

1. IIb positive disease found on clinical exam, CT Scan or intraoperatively (gross appearance or positive margins of frozen section of level IIa)
2. Previous neck RT
3. Previous chemotherapy
4. Invasion of spinal accessory nerve (SAN) by neck malignancy (evident on physical exam, CT scan or intraoperatively (gross appearance).
5. Previous neck dissection
6. Previous SAN injury or dysfunction
7. Preoperative signs or formal diagnosis of myopathy or neuropathy
8. Previous shoulder injury (muscular or bony)
9. Level V neck dissection
10. Recognized intraoperative sectioning of the SAN
11. Unable to provide informed consent
12. Cardiac pacemaker (contra-indication to EMG/Nerve conduction)
13. Radial forearm free flap on dominant arm

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in Neck Dissection Impairment Index (NDII) score from pre- to post-op. | 6 months per patient

SECONDARY OUTCOMES:
Shoulder strength, range of motion and electromyographic (EMG)/nerve conduction testing | 6 months per patients

CONTACTS AND LOCATIONS:
Overall Officials: Hadi R Seikaly, MD, FRCSC, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make data available to others.

REFERENCES:
- [Background] Ambrosch P, Kron M, Pradier O, Steiner W. Efficacy of selective neck dissection: a review of 503 cases of elective and therapeutic treatment of the neck in squamous cell carcinoma of the upper aerodigestive tract. Otolaryngol Head Neck Surg. 2001 Feb;124(2):180-7. doi: 10.1067/mhn.2001.111598. PMID 11226954
- [Background] Cappiello J, Piazza C, Giudice M, De Maria G, Nicolai P. Shoulder disability after different selective neck dissections (levels II-IV versus levels II-V): a comparative study. Laryngoscope. 2005 Feb;115(2):259-63. doi: 10.1097/01.mlg.0000154729.31281.da. PMID 15689746
- [Background] Smith R, Taylor SM, Trites JR, Smith A. Patterns of lymph node metastases to the submuscular recess. J Otolaryngol. 2007 Aug;36(4):203-7. doi: 10.2310/7070.2007.0033. PMID 17942033
- [Background] Silverman DA, El-Hajj M, Strome S, Esclamado RM. Prevalence of nodal metastases in the submuscular recess (level IIb) during selective neck dissection. Arch Otolaryngol Head Neck Surg. 2003 Jul;129(7):724-8. doi: 10.1001/archotol.129.7.724. PMID 12874072
- [Background] Paleri V, Kumar Subramaniam S, Oozeer N, Rees G, Krishnan S. Dissection of the submuscular recess (sublevel IIb) in squamous cell cancer of the upper aerodigestive tract: prospective study and systematic review of the literature. Head Neck. 2008 Feb;30(2):194-200. doi: 10.1002/hed.20682. PMID 17712854
- [Background] Talmi YP, Hoffman HT, Horowitz Z, McCulloch TM, Funk GF, Graham SM, Peleg M, Yahalom R, Teicher S, Kronenberg J. Patterns of metastases to the upper jugular lymph nodes (the "submuscular recess"). Head Neck. 1998 Dec;20(8):682-6. doi: 10.1002/(sici)1097-0347(199812)20:83.0.co;2-j. PMID 9790288
- [Derived] Dziegielewski PT, McNeely ML, Ashworth N, O'Connell DA, Barber B, Courneya KS, Debenham BJ, Seikaly H. 2b or not 2b? Shoulder function after level 2b neck dissection: A double-blind randomized controlled clinical trial. Cancer. 2020 Apr 1;126(7):1492-1501. doi: 10.1002/cncr.32681. Epub 2019 Dec 24. PMID 31873950